CLINICAL TRIAL: NCT03711500
Title: D-serine Augmentation of Neuroplasticity Based Auditory Learning in Schizophrenia
Brief Title: D-serine Augmentation of Neuroplasticity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Joshua Kantrowitz, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7725
Record Dates: First submitted 2018-10-11; First posted 2018-10-18 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: plasticity
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- D-serine 80 mg/kg (Experimental)
  Interventions: Drug: D-serine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- D-serine 100 mg/kg (Experimental)
  Interventions: Drug: D-serine
- D-serine 120 mg/g (Experimental)
  Interventions: Drug: D-serine

INTERVENTIONS:
Drug: D-serine — Subjects will receive three sessions of auditory remediation paired with either D-serine or Placebo in a 4:1 D-serine:placebo ratio. This will be conducted in 3 separate cohorts of D-serine dose 80, 100 and 120 mg/kg, which 15 subjects per cohort (12 active and 3 placebo) per cohort
  Arms: D-serine 100 mg/kg; D-serine 120 mg/g; D-serine 80 mg/kg
Drug: Placebo — Subjects will receive three sessions of auditory remediation paired with either D-serine or Placebo in a 4:1 D-serine:placebo ratio. This will be conducted in 3 separate cohorts of D-serine dose 80, 100 and 120 mg/kg, which 15 subjects per cohort (12 active and 3 placebo) per cohort
  Arms: Placebo

SUMMARY:
Schizophrenia is a major public health problem associated with cognitive deficits, such as short and long term memory, executive functioning, attention and speed of processing that are amongst the strongest predictors of impaired functional outcome. In addition, schizophrenia patients show reduced "plasticity", defined as reduced learning.

D-serine is a naturally occurring activator of the N-methyl-d-aspartate-type glutamate receptors (NMDAR) in the brain, and this project will assess the optimal dose of D-serine treatment over three sessions of a program designed to measure auditory plasticity.

DETAILED DESCRIPTION:
Schizophrenia (Sz) is a major public health problem associated with core cognitive deficits that are amongst the strongest predictors of impaired functional outcome. In addition, Sz patients show reduced cortical neuroplasticity, defined as reduced learning during training on exercises that place implicit, increasing demands on early auditory information processing. As improved auditory processing can facilitate gains in those cognitive processes that are more proximal to daily functioning (e.g., verbal memory, executive functioning), enhancing neuroplasticity for better auditory processing represents an unmet clinical need and a rate-limiting first step prior to remediating cognition and overall function.

As supported by recently published data and review, the study proposes that localized N-methyl-D-aspartate-type glutamate receptor (NMDAR) dysfunction leads to impaired auditory neuroplasticity, which in turn leads to impaired cognition. Over recent years, NMDAR glycine site agonists have increasingly been shown to facilitate neuroplasticity in both Sz and healthy volunteers.

D-serine is a NMDAR modulator that when combined with neuroplasticity-based auditory remediation, leads to highly significant, acute improvement in both auditory plasticity and the early auditory processing measures mismatch negativity (MMN) and theta intertrial coherence (theta). Both MMN and theta-ITC are sensitive measures of functional target engagement of both NMDAR agonism and auditory remediation. In a preliminary study, plasticity correlated with reading and working memory, suggesting plasticity improvements are predictive of functionally relevant outcomes. While D-serine appears to be efficacious for neuroplasticity enhancement and target engagement in a dose dependent manner, the optimal dose remains an open question, as does the ability of combined D-serine + neuroplasticity-based auditory remediation to produce sustained, functional improvement. This study utilizes the Early Stage Testing of Pharmacologic or Device-based Interventions for the Treatment of Mental Disorders (R61/R33): RFA-MH-17-702.

The ultimate goal of this study is to enhance efficacy and efficiency of auditory cognitive remediation by augmenting with D-serine. This study will confirm target engagement, pharmacodynamics, functional relationships and the optimal dose (80 vs.100 vs. 120 mg/kg, IND: 122821) of D-serine treatment combined with 3 sessions of our auditory remediation program. As previously, D-serine will be given 30 minutes before sessions, allowing for auditory remediation during peak serum levels and a pharmacodynamic assessment. Successful completion is defined by ≥moderate effect size change in auditory plasticity, MMN and theta, plus a moderate effect size correlation with functionally relevant cognitive measures ("auditory cognition") without safety issues. Successful completion of this study will pave the way for a larger, definitive study pairing D-serine with auditory remediation or testing alternative dose intervals (1x vs. 2x week). In addition to testing a potentially viable treatment, this project will stimulate industry to utilize this methodology to assess the efficacy of novel NMDAR modulators, using D-serine as a "gold-standard."

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50
2. DSM-V diagnosis of schizophrenia or schizoaffective disorder
3. Willing to provide informed consent
4. Auditory Cognitive impairment demonstrated by:

   a .MCCB composite domain score less than or equal to 0.5 standard deviation below normal (T score less than or equal to 45) b. And at least one of the following:
   * MCCB verbal memory domain score less than or equal to 0.5 standard deviation below normal (T score less than or equal to 45)
   * Tone matching score of less than or equal to 77.7%
5. Clinically stable for 2 months (CGI less than or equal to 4)
6. Moderate or lower cognitive disorganization (PANSS P2 less than or equal to 4)
7. Medically stable for study participation
8. Willing to use qualified methods of contraception for the study duration and up to 2 months after its end
9. Fluent English speaker
10. Normal hearing
11. Visual acuity corrected to 20/30
12. An estimated Glomerular Filtration Rate (GFR) greater than or equal to 60
13. Taking an antipsychotic medication other than clozapine at a stable dose for at least 4 weeks
14. Judged clinically not to be at significant suicide or violence risk

Exclusion Criteria:

1. ECG abnormality that is clinically significant in the context of study participation in the opinion of the study cardiologist
2. Current clozapine use
3. Presence of positive history of unstable significant medical or neurological illness
4. Positive toxicology screen for any substances of abuse
5. Substance use disorder (excluding nicotine) within last 60 days
6. Pregnant women or women of child-bearing potential, who are either not surgically-sterile or for outpatients, using appropriate methods of birth control. Women of childbearing potential must have a negative serum -hCG pregnancy test at every visit.
7. Participation in study of investigational medication/device within 4 weeks
8. Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator Section

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - Nathan Kline Institute, Orangeburg, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Govani V, Shastry AM, Iosifescu DV, Govil P, Mayer MR, Sobeih T, Choo TH, Wall MM, Sehatpour P, Kantrowitz JT. Augmentation of learning in schizophrenia by d-serine and auditory remediation is related to auditory and frontally-generated biomarkers: A randomized, double-blind, placebo-controlled study. Schizophr Res. 2023 Oct;260:205-208. doi: 10.1016/j.schres.2023.08.027. Epub 2023 Sep 11. No abstract available. PMID 37690312
- [Derived] Govani V, Shastry A, Iosifescu D, Govil P, Mayer M, Sobeih T, Choo T, Wall M, Sehatpour P, Kantrowitz J. Augmentation of learning in schizophrenia by D-serine is related to auditory and frontally-generated biomarkers: A randomized, double-blind, placebo-controlled study. Res Sq [Preprint]. 2023 May 19:rs.3.rs-2943290. doi: 10.21203/rs.3.rs-2943290/v1. PMID 37293030
- [Derived] Sehatpour P, Iosifescu DV, De Baun HM, Shope C, Mayer MR, Gangwisch J, Dias E, Sobeih T, Choo TH, Wall MM, Medalia A, Saperstein AM, Kegeles LS, Girgis RR, Carlson M, Kantrowitz JT. Dose-Dependent Augmentation of Neuroplasticity-Based Auditory Learning in Schizophrenia: A Double-Blind, Placebo-Controlled, Randomized, Target Engagement Clinical Trial of the NMDA Glutamate Receptor Agonist d-serine. Biol Psychiatry. 2023 Jul 15;94(2):164-173. doi: 10.1016/j.biopsych.2023.01.015. Epub 2023 Jan 28. PMID 36958998

RESULTS

PARTICIPANT FLOW:
Groups:
- D-serine 80 mg/kg: D-serine 80 m/kg
- D-serine 100 mg/kg: D-serine 100 mg/kg
- D-serine 120 mg/kg: D-serine 120 mg/kg
- Placebo: Placebo
Period: Overall Study
Arm/Group | D-serine 80 mg/kg | D-serine 100 mg/kg | D-serine 120 mg/kg | Placebo
Started | 12 | 12 | 12 | 9
Completed | 12 | 11 (One subject completed 2 of three treatment sessions, with LOCF carried forward for analysis) | 12 | 9
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-serine 80 mg/kg | Placebo | D-serine 100 mg/kg | D-serine 120 mg/g | Total
Number analyzed (Participants) | 12 | 9 | 12 | 12 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (9.6) | 34.8 (8) | 37.6 (6.6) | 35.9 (8.4) | 35.9 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 6 | 0 | 9
  Male | 11 | 7 | 6 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 6 | 3 | 21
  Not Hispanic or Latino | 5 | 4 | 6 | 9 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 9 | 12 | 12 | 45

OUTCOME MEASURES:

1. Primary Outcome: Plasticity Improvement (Change in Tone Matching Threshold)
Description: Participants underwent three treatment sessions, 1x week.
  This is the outcome of the auditory remediation. In Auditory Remediation, participants are presented with paired tones (e.g. Stimulus 1 ("reference") and Stimulus 2 ("test"): S1 and S2) and indicate which tone is higher in pitch (frequency). In the first pair, the ratio is 50% (e.g. 1000±500 Hz). A two-down/one-up staircase procedure is used to adjust the ratio to maintain a steady (~70% correct) level of performance across the trial.
  The tone matching threshold was calculated at the initial plateau (trials 20-30 during treatment session 1) and at the end of treatment session three. Plasticity Improvement was operationalized as change in threshold from initial plateau to the end of treatment visit 3. Larger (more positive) values represent greater improvement in threshold. Zero would represent no improvement. Values were log transformed.
Time Frame: At the end of Treatment session 3 (3rd of three sessions)
Population: randomized
Measure: Mean (Standard Deviation); unit: log ratio
Arm/Group | D-serine 80 mg/kg | Placebo | D-serine 100 mg/kg | D-serine 120 mg/g
Number analyzed (Participants) | 12 | 9 | 12 | 12
log ratio | 13.9 (17.5) | 5.3 (10.8) | 11 (16.4) | -0.05 (14.1)

2. Primary Outcome: Mismatch Negativity (MMN)
Description: MMN is measured by electroencephalogram (EEG). MMN will be obtained independently to pitch stimuli utilizing the same base frequency as the plasticity task described in outcome 1. MMN was assessed immediately before the first dose and immediately after treatment sessions 2 and 3. MMN will be generated using previously published methods. Peak amplitude at frontocentral electrodes within predefined latency range will be primary outcome measure. This value represents the mean MMN to pitch post baseline (after sessions 2 and 3). More negative represents larger MMN.
Time Frame: Post baseline
Population: randomized
Measure: Mean (Standard Deviation); unit: amplitude, micro volts
Arm/Group | D-serine 80 mg/kg | Placebo | D-serine 100 mg/kg | D-serine 120 mg/g
Number analyzed (Participants) | 12 | 9 | 12 | 12
amplitude, micro volts | -1.83 (2.1) | -1.05 (1.6) | -2.71 (1.7) | -0.56 (1.5)

3. Primary Outcome: Theta Intertrial Coherence (Theta)
Description: Theta is measured by EEG, during the motor-preparation interval (200-500 ms post-the second tone: S2) during the auditory remediation task. Theta inter-trial coherence (ITC) reflects the consistency of spectral response across repeated trials ranging from 0 (no consistency) to 1 (perfect consistency). Higher values represent better consistency.
Time Frame: Week 1
Population: randomized
Measure: Mean (Standard Deviation); unit: correlation coefficient (r)
Arm/Group | D-serine 80 mg/kg | Placebo | D-serine 100 mg/kg | D-serine 120 mg/g
Number analyzed (Participants) | 12 | 9 | 12 | 12
correlation coefficient (r) | .229 (.06) | .241 (.06) | 0.274 (.06) | .241 (.07)

4. Primary Outcome: Number of Patients With Granular Casts
Description: This is a safety measure conducted by urinalysis after each D-serine dose. The outcome is the count of participants with granular casts.
Time Frame: Three weeks
Measure: Count of Participants; unit: Participants
Arm/Group | D-serine 80 mg/kg | Placebo | D-serine 100 mg/kg | D-serine 120 mg/g
Number analyzed (Participants) | 12 | 9 | 12 | 12
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | D-serine 80 mg/kg | Placebo | D-serine 100 mg/kg | D-serine 120 mg/g
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03711500/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03711500/SAP_003.pdf